CLINICAL TRIAL: NCT06426771
Title: Investigation of Dietary Inflammatory Index, Dietary Phytochemical Index and NRF Nutrient Density in Patients With High and Low Antimullerian Hormone Levels
Brief Title: Effect of Antimullerian Hormone Levels on the Inflammatory Index, Phytochemical Index and NRF Nutrient Density
Acronym: AMH
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mujde Can Ibanoglu, Assoc. Prof, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: 02/10 28.02.2024
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: AMH; Diet Habit; Ovarian Failure; Polycystic Ovary Syndrome
Keywords: NRF Nutrient Density Index; Dietary Inflammatory Index; Phytochemical Index; anti-Müllerian hormone
MeSH Terms: conditions — Feeding Behavior; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low AMH Levels-: AMH levels: those with low AMH levels (<1.2 ng/ml): 30 participants
  Interventions: Behavioral: Dietary Inflammatory Index; Diagnostic Test: hormone profile
- Normal AMH levels-: normal AMH levels (1.2-3.32 ng/ml): 30 participants
  Interventions: Behavioral: Dietary Inflammatory Index; Diagnostic Test: hormone profile
- High AMH levels-: high AMH levels (>3.32 ng/ml): 30 Participants
  Interventions: Behavioral: Dietary Inflammatory Index; Diagnostic Test: hormone profile

INTERVENTIONS:
Behavioral: Dietary Inflammatory Index — The aim of this study was to compare the dietary habits of patients with PCOS and an AMH value of >3.32 ng/ml, of patients with low ovarian reserve without PCOS and an AMH value of less than 1.2 ng/ml and of patients with normal AMH values (between 1.2-3.32 ng/ml) according to Dietary Nutrient Density according to Dietary Inflammatory Index, Dietary Phytochemical Index and Nutrient Rich Food Index.
  Other Names: Dietary Phytochemical Index; Nutrient Rich Food Index
Diagnostic Test: hormone profile — In the routine practice of the PCOS clinic, about 7 ml of blood is taken in a vacuum gel tube for hormonal and biochemical analysis by medical staff. The blood samples are centrifuged by the researchers at 1000xg for 20 minutes. In the next step, the supernatant part is separated and transferred to 3 mL Ependorfs. These samples are used to determine the levels of anti-Müllerian hormone (AMH), oestradiol, LH and FSH, which are routinely determined at the PCOS clinic.

SUMMARY:
The aim of the study was to calculate the dietary inflammatory index, dietary phytochemical index and NRF nutrient density of the dietary pattern routinely consumed by women and to assess whether there is a difference between PCOS patients with high AMH levels and the group with low AMH levels.

DETAILED DESCRIPTION:
There is currently growing interest in the relationship between lifestyle, reproductive health and fertility. Recent research emphasizes the influence of environmental and lifestyle factors such as stress, diet and nutritional status on reproductive health. Ovarian reserve refers to the number and quality of eggs and is an indicator of reproductive potential. Ovarian reserve is inversely proportional to the chronological age of the mother, which is the most important determinant of reproductive capacity and reproductive success. It has been shown that reproductive aging accelerates after the age of 35. Therefore, the assessment of ovarian reserve is an important step in both the evaluation and treatment of infertility. Markers of ovarian reserve include antral follicle count (AFC), which is determined by transvaginal ultrasound, and serum levels of various biomarkers such as anti-Müllerian hormone (AMH), follicle-stimulating hormone (FSH), luteinizing hormone (LH) and estradiol. Studies show that certain dietary patterns and the intake of certain nutrients are associated with endometriosis, ovarian reserve and egg quality, ovarian infertility and fertility. In addition, there is evidence that modifiable lifestyle factors, such as adherence to certain dietary habits and avoidance of environmental toxins, may also have positive effects on ovarian reserve. Recent studies have shown that women's nutritional status, body mass index and eating habits influence ovarian reserve.

The Dietary Inflammatory Index (DII) is an index developed to assess the impact of general dietary habits on inflammation. It is known that the dietary inflammatory index is high in chronic diseases associated with inflammation. The Phytochemical Index is a calculation based on the consumption of fruits high in phytochemicals, all vegetables except potatoes, legumes, whole grains and whole grain-containing foods, and oilseeds that provides information about the level of phytochemicals in the diet. The NRF Nutrient Density Index is a continuous function and represents an arithmetic combination of weighted variables. In this continuous function algorithm, the negative part (foods that should be restricted) is subtracted from the positive part (foods that should be consumed). In the calculation phase of this model, foods were scored according to their nutrient content per 100 kcal and per serving size. By calculating the nutrient density of the food consumed, the quality of the person's diet can be determined.

Based on this information, it was planned to compare these 3 nutritional indices in patients diagnosed with PCOS with an AMH level above 3.32 ng/ml, in the low ovarian reserve group without a PCOS diagnosis with an AMH level below 1.2 ng/ml and in normo-responder patients with an AMH level between these two values.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40,
* No underlying metabolic disease (type 2 diabetes, hypertension, diagnosed anemia),
* Female patients with AMH levels in our hospital,
* Participants attending the PCOS clinic and under the care of our hospital dietitian will be enrolled in the study.

Exclusion Criteria:

1. Age < 18 and > 40 years;
2. Menopause, pregnancy or breastfeeding in the last 6 months;
3. Hyperandrogenism and/or biochemical hyperandrogenemia due to secondary causes, including congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome, hyperprolactinemia, thyroid dysfunction, and adrenal disease),
4. Pre-existing systemic or psychiatric illnesses
5. Taking medication that affects carbohydrate or fat metabolism (contraceptive pills, metformin, antiepileptic drugs, antipsychotics, statins and fish oil);
6. Certain nutritional therapies or hypocaloric diet in the last three months; supplementation with antioxidants, vitamins or minerals;
7. Taking medications that can affect fluid balance, such as non-steroidal anti-inflammatory drugs, diuretics, etc.
8. Female patients with implanted pacemakers or defibrillators due to the theoretical possibility of impaired device activity.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was designed as a cross-sectional cohort study including individuals who were followed up in the PCOS Clinic and dietetic department of Etlik Zübeyde Hanım Gynaecology Training and Research Hospital. Patients will be divided into 3 groups according to AMH value as those with low AMH value, those with normal AMH value and those with high AMH value (11).
  The study will include 90 individuals who agreed to be included in the study and accepted the consent form verbally and in writing.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
AMH levels according to dietary indexes | 6 months
  Patients with low, normal and high AMH values are examined for differences in the indices calculated according to nutrient density.

CONTACTS AND LOCATIONS:
Overall Officials: Mujde Can Ibanoglu, Principal Investigator — Ankara Etlik Zubeyde Hanım Women's Health Training and Research Hospital, Ankara, Turkey.
Locations (1):
- Etlik Zübeyde Hanım, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lakoma K, Kukharuk O, Sliz D. The Influence of Metabolic Factors and Diet on Fertility. Nutrients. 2023 Feb 27;15(5):1180. doi: 10.3390/nu15051180. PMID 36904180
- [Result] Barrea L, Arnone A, Annunziata G, Muscogiuri G, Laudisio D, Salzano C, Pugliese G, Colao A, Savastano S. Adherence to the Mediterranean Diet, Dietary Patterns and Body Composition in Women with Polycystic Ovary Syndrome (PCOS). Nutrients. 2019 Sep 23;11(10):2278. doi: 10.3390/nu11102278. PMID 31547562